CLINICAL TRIAL: NCT03100344
Title: Randomized, Double-blind, Multi-center, Parallel-group, Placebo-controlled Dose-ranging Study to Assess the Efficacy and Safety of Nemolizumab in Moderate-to-severe Atopic Dermatitis Subjects With Severe Pruritus Receiving Topical Corticosteroids (TCS)
Brief Title: Dose-ranging Study of Nemolizumab in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.03.SPR.114322
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Nemolizumab (low dose)
  Interventions: Drug: Nemolizumab
- Group 2 (Experimental): Nemolizumab (medium dose)
  Interventions: Drug: Nemolizumab
- Group 3 (Experimental): Nemolizumab (high dose)
  Interventions: Drug: Nemolizumab
- Group 4 (Placebo Comparator): Nemolizumab placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Injection every 4 weeks during 24 weeks (last injection at week 20)
  Arms: Group 1; Group 2; Group 3
Drug: Placebo — Injection every 4 weeks during 24 weeks (last injection at week 20)
  Arms: Group 4

SUMMARY:
Assess the efficacy of several subcutaneous doses of nemolizumab in moderate-to-severe atopic dermatitis (AD) subjects with severe pruritus receiving TCS, who were not adequately controlled with topical treatments.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of several subcutaneous doses of nemolizumab in moderate-to-severe atopic dermatitis (AD) subjects with severe pruritus receiving topical corticosteroids, who were not adequately controlled with topical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years (or legal age when higher)
* Chronic AD, that has been present for at least 2 years before the visit
* Eczema Area and Severity Index (EASI) score ≥12
* Investigator Global Assessment (IGA) score ≥ 3
* AD involvement ≥ 10% of Body Surface Area (BSA)
* Severe pruritus on at least 3 of the last 7 days before the visit
* Documented recent history (within 6 months before the visit) of inadequate response to topical medications
* Female subjects must fulfill one of the criteria below:

  * Female subjects of non-childbearing potential
  * Female subjects of childbearing potential who agree to a true abstinence or to use an effective or highly effective method of contraception throughout the clinical trial and for 120 days after the last study drug administration

Exclusion Criteria:

* Body weight < 45 kg
* subjects with a medical history of asthma requiring hospitalization in the last 12 months before screening visit and/or whose asthma has not been well-controlled during the last 3 months before the screening visit and/or Peak Expiratory Flow (PEF) <80% of the predicted value
* Cutaneous bacterial or viral infection within 1 week before the screening visit or during the run-in period
* Infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 1 week before the screening visit or during the run-in period
* History of intolerance to low or mid potency TCS or for whom TCS is not advisable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (26):
  - Galderma Investigational site, Birmingham, Alabama
  - Galderma Investigational site, Fort Smith, Arkansas
  - Galderma Investigational site, Beverly Hills, California
  - Galderma Investigational site, Fountain Valley, California
  - Galderma Investigational site, Fremont, California
  - Galderma Investigational site, Rolling Hills Estates, California
  - Galderma Investigational site, Santa Ana, California
  - Galderma Investigational site, Santa Monica, California
  - Galderma Investigational site, Miami, Florida
  - Galderma Investigational site, Tampa, Florida
  - Galderma Investigational Site, Tampa, Florida
  - Galderma Investigational site, Columbus, Georgia
  - Galderma Investigational site, Sandy Springs, Georgia
  - Galderma Investigational Site, Darien, Illinois
  - Galderma Investigational Site, Overland Park, Kansas
  - Galderma Investigational site, New Orleans, Louisiana
  - Galderma Investigational Site, Farmington Hills, Michigan
  - Galderma Investigational site, Forest Hills, New York
  - Galderma Investigational site, New York, New York
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational site, Chapel Hill, North Carolina
  - Galderma Investigational Site, Johnston, Rhode Island
  - Galderma Investigational site, Dallas, Texas
  - Galderma Investigational site, San Antonio, Texas
  - Galderma Investigational Site, Waco, Texas
  - Galderma Investigational site, Richmond, Virginia
- Australia (4):
  - Galderma Investigational Site, Benowa
  - Galderma Investigational Site, Kogarah
  - Galderma Investigational Site, Melbourne
  - Galderma Investigational Site, Phillip
- Canada (8):
  - Galderma Investigational Site, Calgary
  - Galderma Investigational Site, Markham
  - Galderma Investigational Site, Oakville
  - Galderma Investigational Site, Ottawa
  - Galderma Investigational Site, Peterborough
  - Galderma Investigational Site, Richmond Hill
  - Galderma Investigational Site, Sainte-Foy
  - Galderma Investigational Site, Waterloo
- France (6):
  - Galderma Investigational Site, Bordeaux
  - Galderma Investigational Site, Lille
  - Galderma Investigational Site, Marseille
  - Galderma Investigational Site, Nice
  - Galderma Investigational Site, Paris
  - Galderma Investigational Site, Toulouse
- Germany (12):
  - Galderma Investigational Site, Berlin
  - Galderma Investigational Site, Darmstadt
  - Galderma Investigational Site, Erlangen
  - Galderma Investigational Site, Frankfurt
  - Galderma Investigational Site, Hamburg
  - Galderma Investigational Site, Hannover
  - Galderma Investigational Site, Heidelberg
  - Galderma Investigational Site, Langenau
  - Galderma Investigational Site, Mainz
  - Galderma Investigational Site, München
  - Galderma Investigational Site, Osnabrück
  - Galderma Investigational Site, Stuttgart
- Poland (6):
  - Galderma Investigational Site, Katowice
  - Galderma Investigational Site, Krakow
  - Galderma Investigational Site, Lodz
  - Galderma Investigational Site, Lublin
  - Galderma Investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw

REFERENCES:
- [Derived] Silverberg JI, Pinter A, Pulka G, Poulin Y, Bouaziz JD, Wollenberg A, Murrell DF, Alexis A, Lindsey L, Ahmad F, Piketty C, Clucas A. Phase 2B randomized study of nemolizumab in adults with moderate-to-severe atopic dermatitis and severe pruritus. J Allergy Clin Immunol. 2020 Jan;145(1):173-182. doi: 10.1016/j.jaci.2019.08.013. Epub 2019 Aug 23. PMID 31449914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 57 investigational sites in Australia, Canada, Germany, France, Poland and the United States.
Pre-assignment Details: In this study, 226 participants with moderate-to-severe atopic dermatitis (AD) were randomized across the 4 treatment groups after a 2 to 4-week run-in period. All participants underwent inclusion and exclusion criteria assessment and all eligible participants signed the informed consent before undergoing any study related procedures.
Groups:
- Placebo: Randomized participants received Nemolizumab placebo subcutaneous injection every 4 weeks during 24 week treatment period (last injection at Week 20). As background therapy a medium potency topical corticosteroids (TCS) (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
- Nemolizumab (10 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at Week 20) with a loading dose of 20mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
- Nemolizumab (30 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at Week 20) with a loading dose of 60mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
- Nemolizumab (90 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at Week 20). As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
Period: Overall Study
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Started | 57 | 55 | 57 | 57
Completed | 43 | 44 | 50 | 45
Not Completed | 14 | 11 | 7 | 12
Not completed — Adverse Event | 0 | 3 | 2 | 3
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 7 | 4 | 8
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants. The ITT population was analyzed according to the treatment groups or stratum assigned at randomization.
Groups:
- Placebo: Randomized participants received Nemolizumab placebo subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20). As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) for areas where medium potency TCS are considered unsafe.
- Nemolizumab (10 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 weeks treatment period (last injection at week 20) with a loading dose of 20 mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) for areas where medium potency TCS are considered unsafe.
- Nemolizumab (30 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20) with a loading dose of 60 mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) for areas where medium potency TCS are considered unsafe.
- Nemolizumab (90 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20). As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) for areas where medium potency TCS are considered unsafe.
- Total: Total of all reporting groups
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg) | Total
Number analyzed (Participants) | 57 | 55 | 57 | 57 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 53 | 51 | 51 | 209
  >=65 years | 3 | 2 | 6 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.01) | 35.3 (14.83) | 40.2 (16.64) | 40.9 (14.95) | 39.3 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 28 | 31 | 111
  Male | 31 | 29 | 29 | 26 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 4 | 11 | 6 | 4 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 3 | 10 | 8 | 29
  White | 45 | 38 | 40 | 44 | 167
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 4
Height [Mean (Standard Deviation); unit: centimetre] | 170.0 (10.28) | 169.7 (8.98) | 171.5 (8.55) | 170.6 (9.94) | 170.5 (9.43)
Weight [Mean (Standard Deviation); unit: kilogram] | 80.58 (18.835) | 73.72 (14.629) | 76.90 (18.613) | 80.49 (22.770) | 77.96 (19.052)
Body mass index [Mean (Standard Deviation); unit: kilogram per square metre] | 27.79 (5.638) | 25.54 (4.429) | 26.18 (6.370) | 27.51 (6.694) | 26.77 (5.894)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) at Week 24
Description: EASI is a composite score ranging from 0 to 72.The severity of erythema, induration/papulation, excoriation, and lichenification was assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. Higher scores indicate worse outcome.
Time Frame: From Baseline to Week 24
Population: All participants in intent-to-treat (ITT) population who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Placebo: Randomized participants received Nemolizumab placebo subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20). As background therapy , a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe
- Nemolizumab (10 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20) with a loading dose of 20 mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
- Nemolizumab (30 mg): Randomized participants received Nemolizumab subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20) with a loading dose of 60 mg. As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
percentage change | -58.4 (31.99) | -72.2 (25.96) | -73.4 (29.67) | -69.2 (31.06)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Other — mixed-effect model for repeated measures (MMRM); p = 0.051, Kenward-Rogers; mean difference of percentage changes = -13.6, 95% CI 2-sided [-27.3 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Other — mixed-effect model for repeated measures (MMRM); p = 0.016, Kenward Roger; mean difference of percentage changes = -16.7, 95% CI 2-sided [-30.2 to -3.2]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Other — mixed-effect model for repeated measures (MMRM); p = 0.322, Kenward Roger; mean difference of percentage changes = -6.8, 95% CI 2-sided [-20.5 to 6.8]

2. Secondary Outcome: Number of Participants Achieving Pruritus Categorical Scale (PCS) Success (Defined as a Weekly Prorated Rounded Average PCS ≤1 [None - Mild]) at Week 24
Description: The 4-point pruritus categorical scale was provided in their local language for the participants to report the intensity of their pruritus. Overall itching was scored as 0 for absence of pruritus and 3 for severe pruritus (bothersome itching/scratching that disturbs sleep). Higher scores indicate worse outcome.
Time Frame: Week 24
Population: ITT population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Randomized participants received Nemolizumab placebo subcutaneous injection every 4 weeks during 24 week treatment period (last injection at week 20). As background therapy a medium potency TCS (mometasone furoate 0.1% cream or hydrocortisone butyrate 0.1% cream) was used for the body and a low potency TCS (hydrocortisone acetate 0.05-1% cream or desonide 0.05% cream) was used for areas where medium potency TCS are considered unsafe.
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants | 13 | 23 | 31 | 20
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.9, 95% CI 2-sided [2.0 to 35.8]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 31.4, 95% CI 2-sided [14.7 to 48.2]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Superiority; p = 0.154, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-4.2 to 28.6]

3. Secondary Outcome: Number of Participants With an Improvement of Weekly Average Peak Pruritus Numeric Rating Scale (NRS) ≥4 at Each Timepoint up to Week 24
Description: Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Time Frame: From Week 1 to Week 24
Population: ITT population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1: number analyzed (Participants) | 55 | 52 | 53 | 52
  Week 1 | 3 | 9 | 10 | 6
  Week 2: number analyzed (Participants) | 53 | 50 | 55 | 50
  Week 2 | 6 | 19 | 21 | 17
  Week 4: number analyzed (Participants) | 52 | 50 | 51 | 49
  Week 4 | 4 | 19 | 27 | 22
  Week 8: number analyzed (Participants) | 50 | 45 | 51 | 46
  Week 8 | 11 | 22 | 36 | 26
  Week 12: number analyzed (Participants) | 41 | 41 | 48 | 42
  Week 12 | 13 | 26 | 38 | 24
  Week 16: number analyzed (Participants) | 39 | 39 | 47 | 40
  Week 16 | 12 | 30 | 39 | 25
  Week 20: number analyzed (Participants) | 34 | 37 | 41 | 36
  Week 20 | 13 | 27 | 34 | 27
  Week 24: number analyzed (Participants) | 32 | 33 | 36 | 31
  Week 24 | 14 | 25 | 28 | 24
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.062, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.9, 95% CI 2-sided [-0.4 to 22.2]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p = 0.042, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [0.8 to 23.6]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.307, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-4.7 to 15.0]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.0, 95% CI 2-sided [9.3 to 38.7]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.2, 95% CI 2-sided [11.4 to 40.9]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.0, 95% CI 2-sided [4.9 to 33.1]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 27.6, 95% CI 2-sided [13.5 to 41.7]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 40.3, 95% CI 2-sided [25.7 to 54.8]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 31.6, 95% CI 2-sided [17.4 to 45.8]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [4.2 to 37.1]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p < 0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 43.7, 95% CI 2-sided [27.6 to 59.9]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.1, 95% CI 2-sided [9.7 to 42.6]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.4, 95% CI 2-sided [7.3 to 41.4]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 43.6, 95% CI 2-sided [27.4 to 59.9]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.1, 95% CI 2-sided [2.4 to 35.9]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 33.3, 95% CI 2-sided [16.4 to 50.2]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 47.2, 95% CI 2-sided [31.2 to 63.2]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.010, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.8, 95% CI 2-sided [6.1 to 39.4]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.3, 95% CI 2-sided [9.2 to 43.5]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 36.7, 95% CI 2-sided [20.1 to 53.3]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.5, 95% CI 2-sided [7.6 to 41.4]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [3.6 to 38.1]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.3, 95% CI 2-sided [7.4 to 41.3]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.050, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [0.4 to 34.4]

4. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 24
Description: SCORAD ranges from 0 to 103 and has three components: extent (body surface area [BSA]), signs, and symptoms of AD. The severity of the 6 signs of AD (erythema/darkening, edema/papulation, oozing/crusting, excoriation, lichenification/prurigo and dryness), was assessed, each on a scale ranging from 0 (none) to 3 (severe).The component of extent corresponded to the extent of BSA affected by atopic dermatitis.The BSA involvement of AD was assessed for each part of the body (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]), and was reported as a percentage of all major body sections combined. Participants were also asked to evaluate their symptoms of pruritus and sleep loss (average for the last 3 days/nights), each evaluated on a Visual analog scale (VAS) from 0 to 10. Higher scores indicate worse outcome.
Time Frame: Baseline, Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Percentage change | -42.6 (28.25) | -60.8 (25.04) | -62.5 (25.37) | -55.9 (25.85)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Other — mixed-effect model for repeated measures; p = 0.017, Kenward Roger; mean difference of percentage changes = -14.4, 95% CI 2-sided [-26.2 to -2.7]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Other — mixed-effect model for repeated measures; p = 0.058, Kenward Roger; mean difference of percentage changes = -11.3, 95% CI 2-sided [-23.1 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of percentage changes = -20.0, 95% CI 2-sided [-31.6 to -8.3]

5. Secondary Outcome: Absolute Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
units on a scale | -27.9 (19.61) | -40.1 (19.19) | -40.6 (17.22) | -36.1 (16.56)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Other — mixed-effect model for repeated measures; p = 0.016, Kenward Roger; mean difference of absolute changes = -9.6, 95% CI 2-sided [-17.5 to -1.8]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Other — mixed-effect model for repeated measures; p = 0.001, Kenward Roger; mean difference of absolute changes = -12.8, 95% CI 2-sided [-20.6 to -5.1]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Other — mixed-effect model for repeated measures; p = 0.058, Kenward Roger; mean difference of absolute changes = -7.6, 95% CI 2-sided [-15.4 to 0.3]

6. Secondary Outcome: Percent Change From Baseline in Weekly Average Sleep Disturbance Numeric Rating Scale (NRS) at Week 24
Description: The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants were asked the following questions in their local language: how would you rate your sleep last night?: On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Time Frame: Baseline, Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Percentage change | -50.7 (33.52) | -75.4 (27.64) | -76.2 (23.60) | -74.9 (29.39)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of percentage changes = -24.5, 95% CI 2-sided [-37.8 to -11.2]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of percentage changes = -31.7, 95% CI 2-sided [-44.9 to -18.6]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of percentage changes = -25.1, 95% CI 2-sided [-38.4 to -11.8]

7. Secondary Outcome: Absolute Change From Baseline in Weekly Average Sleep Disturbance Numeric Rating Scale (NRS) at Week 24
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
units on a scale | -3.9 (2.74) | -6.2 (2.34) | -5.7 (2.51) | -5.8 (2.62)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of absolute changes = -2.0, 95% CI 2-sided [-3.1 to -1.0]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of absolute changes = -2.3, 95% CI 2-sided [-3.4 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Test type: Other — mixed-effect model for repeated measures; p < 0.001, Kenward Roger; mean difference of absolute changes = -1.9, 95% CI 2-sided [-3.0 to -0.9]

8. Secondary Outcome: Number of Participants Achieving Investigator's Global Assessment (IGA) Success (Defined as IGA 0 [Clear] or 1 [Almost Clear]) at Each Timepoint up to Week 24
Description: IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used to evaluate the global severity of AD. Higher scores indicate worse outcome.
Time Frame: From Week 1 to Week 24
Population: ITT population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1: number analyzed (Participants) | 55 | 53 | 55 | 57
  Week 1 | 1 | 1 | 2 | 0
  Week 2: number analyzed (Participants) | 55 | 55 | 55 | 57
  Week 2 | 2 | 1 | 4 | 1
  Week 4: number analyzed (Participants) | 54 | 55 | 54 | 56
  Week 4 | 2 | 1 | 9 | 7
  Week 8: number analyzed (Participants) | 52 | 53 | 52 | 54
  Week 8 | 2 | 3 | 10 | 11
  Week 12: number analyzed (Participants) | 45 | 46 | 50 | 51
  Week 12 | 6 | 6 | 15 | 15
  Week 16: number analyzed (Participants) | 44 | 46 | 47 | 45
  Week 16 | 7 | 9 | 19 | 15
  Week 20: number analyzed (Participants) | 39 | 42 | 46 | 41
  Week 20 | 9 | 11 | 19 | 14
  Week 24: number analyzed (Participants) | 38 | 40 | 44 | 40
  Week 24 | 12 | 14 | 21 | 13
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); At week 1; Test type: Other; p = 0.970, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-4.9 to 5.1]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); At week 1; Test type: Other; p = 0.574, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-4.1 to 7.5]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); At week 1; Test type: Other; p = 0.311, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.2 to 1.7]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); At week 24; Test type: Other; p = 0.598, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-11.3 to 19.8]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); At week 24; Test type: Other; p = 0.066, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.5, 95% CI 2-sided [-0.4 to 31.4]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); At week 24; Test type: Other; p = 0.826, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-13.5 to 16.9]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.558, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.7 to 4.1]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.413, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-4.7 to 11.6]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.543, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.7 to 4.0]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.583, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-7.6 to 4.2]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.028, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [1.8 to 22.5]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.087, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [-0.9 to 18.3]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.632, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-5.6 to 9.4]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [3.1 to 24.8]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.8, 95% CI 2-sided [4.5 to 27.0]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.974, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-11.2 to 11.6]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p = 0.031, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [1.8 to 29.3]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.9, 95% CI 2-sided [-0.3 to 28.2]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.553, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-9.0 to 16.9]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [6.1 to 35.8]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.061, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.9, 95% CI 2-sided [-0.3 to 28.2]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.585, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-10.1 to 18.0]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [2.0 to 32.8]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.254, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [-5.9 to 23.1]

9. Secondary Outcome: Number of Participants With Eczema Area and Severity Index (EASI)-50 (Defined as Achieving 50% Reduction From Baseline in EASI Score) at Each Visit up to Week 24
Description: EASI is a composite score ranging from 0 to 72. The severity of erythema, induration/papulation, excoriation, and lichenification were assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. Higher scores indicate worse outcome.
Time Frame: From Week 1 to Week 24
Population: ITT Population:All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1: number analyzed (Participants) | 55 | 53 | 55 | 57
  Week 1 | 4 | 6 | 12 | 11
  Week 2: number analyzed (Participants) | 55 | 55 | 55 | 57
  Week 2 | 8 | 18 | 18 | 21
  Week 4: number analyzed (Participants) | 54 | 55 | 54 | 56
  Week 4 | 14 | 22 | 29 | 24
  Week 8: number analyzed (Participants) | 52 | 53 | 52 | 54
  Week 8 | 15 | 26 | 31 | 31
  Week 12: number analyzed (Participants) | 45 | 46 | 50 | 51
  Week 12 | 20 | 30 | 36 | 30
  Week 16: number analyzed (Participants) | 44 | 46 | 47 | 45
  Week 16 | 21 | 30 | 34 | 32
  Week 20: number analyzed (Participants) | 39 | 42 | 46 | 41
  Week 20 | 23 | 32 | 38 | 33
  Week 24: number analyzed (Participants) | 38 | 40 | 44 | 40
  Week 24 | 25 | 33 | 38 | 31
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.487, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-6.8 to 14.3]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [1.6 to 26.5]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.053, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.0, 95% CI 2-sided [0.2 to 23.8]
Statistical Analysis 4: Comparison: Placebo; Week 2; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.5, 95% CI 2-sided [3.2 to 33.8]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.027, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [2.4 to 32.3]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.7, 95% CI 2-sided [7.3 to 38.1]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.086, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.2, 95% CI 2-sided [-1.7 to 32.2]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.2, 95% CI 2-sided [9.3 to 43.1]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.050, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.3, 95% CI 2-sided [0.5 to 34.2]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [3.3 to 38.1]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 27.9, 95% CI 2-sided [10.7 to 45.0]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 27.9, 95% CI 2-sided [10.7 to 45.0]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.041, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.3, 95% CI 2-sided [1.3 to 37.3]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 27.9, 95% CI 2-sided [10.4 to 45.4]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.063, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.3, 95% CI 2-sided [-0.5 to 35.2]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.064, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.6, 95% CI 2-sided [-0.4 to 35.6]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.6, 95% CI 2-sided [4.9 to 40.3]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.041, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.1, 95% CI 2-sided [1.3 to 36.9]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.064, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.6, 95% CI 2-sided [-0.4 to 35.6]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.0, 95% CI 2-sided [8.6 to 43.4]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.064, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.2, 95% CI 2-sided [-0.6 to 35.0]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.094, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.9, 95% CI 2-sided [-2.0 to 33.8]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.4, 95% CI 2-sided [5.1 to 39.6]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.273, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.2, 95% CI 2-sided [-7.7 to 28.0]

10. Secondary Outcome: Number of Participants With Eczema Area and Severity Index (EASI)-75 (Defined as Achieving 75% Reduction From Baseline in EASI Score) at Each Visit up to Week 24
Description: EASI is a composite score ranging from 0 to 72.The severity of erythema, induration/papulation, excoriation, and lichenification were assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. Higher scores indicate worse outcome.
Time Frame: From Week 1 to Week 24
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1: number analyzed (Participants) | 55 | 53 | 55 | 57
  Week 1 | 2 | 2 | 3 | 3
  Week 2: number analyzed (Participants) | 55 | 55 | 55 | 57
  Week 2 | 4 | 5 | 6 | 12
  Week 4: number analyzed (Participants) | 54 | 55 | 54 | 56
  Week 4 | 3 | 7 | 12 | 15
  Week 8: number analyzed (Participants) | 52 | 53 | 52 | 54
  Week 8 | 7 | 10 | 21 | 15
  Week 12: number analyzed (Participants) | 45 | 46 | 50 | 51
  Week 12 | 10 | 15 | 25 | 21
  Week 16: number analyzed (Participants) | 44 | 46 | 47 | 45
  Week 16 | 11 | 18 | 28 | 21
  Week 20: number analyzed (Participants) | 39 | 42 | 46 | 41
  Week 20 | 16 | 21 | 25 | 21
  Week 24: number analyzed (Participants) | 38 | 40 | 44 | 40
  Week 24 | 15 | 20 | 26 | 25
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.979, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-6.8 to 7.0]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p = 0.668, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-5.8 to 9.0]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.658, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-5.8 to 9.2]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.690, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-8.0 to 12.2]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.521, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-6.9 to 13.7]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [1.5 to 26.5]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.172, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-3.1 to 18.0]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.7, 95% CI 2-sided [3.7 to 27.7]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 21.0, 95% CI 2-sided [8.2 to 33.9]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.404, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-7.5 to 18.8]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.5, 95% CI 2-sided [9.4 to 39.6]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.059, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.1, 95% CI 2-sided [-0.1 to 28.2]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.222, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [-5.6 to 25.0]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 26.1, 95% CI 2-sided [10.0 to 42.3]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.22, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.1, 95% CI 2-sided [3.3 to 35.0]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.111, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.3, 95% CI 2-sided [-2.8 to 29.3]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 29.6, 95% CI 2-sided [13.2 to 46.0]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [1.3 to 33.6]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.262, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [-7.3 to 27.4]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.327, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [-8.4 to 25.7]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.083, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.7, 95% CI 2-sided [-1.7 to 33.1]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.255, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [-7.0 to 27.2]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.0, 95% CI 2-sided [2.2 to 35.9]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.053, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [0.3 to 34.6]

11. Secondary Outcome: Number of Participants With Eczema Area and Severity Index (EASI)-90 (Defined as Achieving 90% Reduction From Baseline in EASI Score) at Each Visit up to Week 24
Description: as for outcome 10
Time Frame: From Week 1 to Week 24
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1: number analyzed (Participants) | 55 | 53 | 55 | 57
  Week 1 | 1 | 1 | 2 | 1
  Week 2: number analyzed (Participants) | 55 | 55 | 55 | 57
  Week 2 | 2 | 0 | 2 | 2
  Week 4: number analyzed (Participants) | 54 | 55 | 54 | 56
  Week 4 | 2 | 1 | 4 | 3
  Week 8: number analyzed (Participants) | 52 | 53 | 52 | 54
  Week 8 | 1 | 3 | 11 | 6
  Week 12: number analyzed (Participants) | 45 | 46 | 50 | 51
  Week 12 | 4 | 7 | 13 | 14
  Week 16: number analyzed (Participants) | 44 | 46 | 47 | 45
  Week 16 | 5 | 10 | 19 | 12
  Week 20: number analyzed (Participants) | 39 | 42 | 46 | 41
  Week 20 | 6 | 13 | 18 | 14
  Week 24: number analyzed (Participants) | 38 | 40 | 44 | 40
  Week 24 | 6 | 13 | 17 | 13
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.970, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-4.9 to 5.1]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p = 0.574, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-4.1 to 7.5]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.985, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-4.8 to 4.8]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.154, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-8.4 to 1.2]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.978, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-6.8 to 6.6]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.978, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-6.8 to 6.6]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.602, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-7.5 to 4.3]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.413, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-4.5 to 11.4]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.658, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-5.7 to 9.1]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.307, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-3.2 to 10.3]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.3, 95% CI 2-sided [6.9 to 27.8]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [0.1 to 17.4]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.325, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-5.4 to 16.5]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [3.1 to 28.1]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.5, 95% CI 2-sided [4.5 to 30.5]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.153, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 9.2, 95% CI 2-sided [-3.2 to 21.7]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 24.4, 95% CI 2-sided [10.3 to 38.4]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-0.7 to 25.1]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.070, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.9, 95% CI 2-sided [-0.8 to 26.6]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [6.5 to 35.3]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.052, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [0.3 to 27.7]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.8, 95% CI 2-sided [-0.7 to 26.3]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.1, 95% CI 2-sided [4.9 to 33.3]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.083, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-1.3 to 25.7]

12. Secondary Outcome: Number of Participants Achieving Investigator Global Assessment (IGA) Success (Defined as IGA 0 [Clear] or 1 [Almost Clear]) and a Reduction of ≥2 Points at Each Visit up to Week 24
Description: as for outcome 8
Time Frame: Week 1 to Week 24
Population: All participants in ITT population who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Participants
  Week 1 | 1 | 1 | 2 | 0
  Week 2 | 2 | 1 | 4 | 1
  Week 4 | 2 | 1 | 9 | 7
  Week 8 | 2 | 3 | 10 | 11
  Week 12 | 6 | 6 | 15 | 15
  Week 16 | 7 | 9 | 19 | 15
  Week 20 | 9 | 11 | 19 | 14
  Week 24 | 12 | 14 | 21 | 13
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.970, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-4.9 to 5.1]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p = 0.574, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-4.1 to 7.5]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.311, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.2 to 1.7]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.558, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.7 to 4.1]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.413, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-4.7 to 11.6]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.543, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.7 to 4.0]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.583, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-7.6 to 4.2]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.028, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [1.8 to 22.5]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.087, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [-0.9 to 18.3]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.632, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-5.6 to 9.4]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [3.1 to 24.8]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.8, 95% CI 2-sided [4.5 to 27.0]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.974, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-11.2 to 11.6]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p = 0.031, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [1.8 to 29.3]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [1.8 to 29.5]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.553, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-9.0 to 16.9]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [6.1 to 35.8]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.061, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.9, 95% CI 2-sided [-0.3 to 28.2]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.585, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-10.1 to 18.0]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [2.0 to 32.8]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.254, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [-5.9 to 23.1]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.598, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-11.3 to 19.8]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.066, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.5, 95% CI 2-sided [-0.4 to 31.4]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.826, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-13.5 to 16.9]

13. Secondary Outcome: Percentage Change From Baseline in Eczema Area and Severity Index (EASI) at Each Visit up to Week 24
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Percentage of change
  Week 1: number analyzed (Participants) | 55 | 53 | 55 | 57
  Week 1 | -12.4 (24.32) | -22.7 (23.54) | -29.3 (31.44) | -28.6 (25.52)
  Week 2: number analyzed (Participants) | 55 | 55 | 55 | 57
  Week 2 | -24.8 (29.16) | -34.9 (27.70) | -40.1 (26.96) | -40.1 (32.83)
  Week 4: number analyzed (Participants) | 54 | 55 | 54 | 56
  Week 4 | -26.5 (33.45) | -40.3 (28.36) | -46.7 (38.49) | -41.8 (41.57)
  Week 8: number analyzed (Participants) | 52 | 53 | 52 | 54
  Week 8 | -28.6 (36.85) | -42.0 (38.15) | -51.7 (47.73) | -49.9 (37.21)
  Week 12: number analyzed (Participants) | 45 | 46 | 50 | 51
  Week 12 | -43.3 (35.22) | -58.5 (28.16) | -64.1 (33.92) | -56.7 (37.25)
  Week 16: number analyzed (Participants) | 44 | 46 | 47 | 45
  Week 16 | -47.6 (32.09) | -59.1 (33.09) | -72.2 (27.59) | -61.8 (41.62)
  Week 20: number analyzed (Participants) | 39 | 42 | 46 | 41
  Week 20 | -57.3 (31.66) | -67.2 (35.18) | -71.6 (29.39) | -70.9 (27.07)
  Week 24: number analyzed (Participants) | 38 | 40 | 44 | 40
  Week 24 | -58.4 (31.99) | -72.2 (25.96) | -73.4 (29.67) | -69.2 (31.06)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.049, Kenward-Rogers; mean difference of percentage changes = -10.0, 95% CI 2-sided [-20.0 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -16.9, 95% CI 2-sided [-26.7 to -7.0]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.002, Kenward Roger; mean difference of percentage changes = -15.7, 95% CI 2-sided [-25.6 to -5.8]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p = 0.084, Kenward Roger; mean difference of percentage changes = -9.8, 95% CI 2-sided [-20.9 to 1.3]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p = 0.004, Kenward Roger; mean difference of percentage changes = -16.2, 95% CI 2-sided [-27.2 to -5.2]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p = 0.008, Kenward Roger; mean difference of percentage changes = -14.8, 95% CI 2-sided [-25.8 to -3.8]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p = 0.044, Kenward Roger; mean difference of percentage changes = -14.0, 95% CI 2-sided [-27.5 to -0.4]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p = 0.002, Kenward Roger; mean difference of percentage changes = -21.1, 95% CI 2-sided [-34.7 to -7.6]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p = 0.026, Kenward Roger; mean difference of percentage changes = -15.3, 95% CI 2-sided [-28.8 to -1.8]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p = 0.062, Kenward Roger; mean difference of percentage changes = -14.8, 95% CI 2-sided [-30.2 to 0.7]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p = 0.003, Kenward Roger; mean difference of percentage changes = -23.4, 95% CI 2-sided [-38.9 to -7.9]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p = 0.009, Kenward Roger; mean difference of percentage changes = -20.6, 95% CI 2-sided [-36.0 to -5.2]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p = 0.022, Kenward Roger; mean difference of percentage changes = -15.9, 95% CI 2-sided [-29.4 to -2.3]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -23.7, 95% CI 2-sided [-37.1 to -10.2]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p = 0.032, Kenward Roger; mean difference of percentage changes = -14.7, 95% CI 2-sided [-28.1 to -1.3]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p = 0.070, Kenward Roger; mean difference of percentage changes = -13.7, 95% CI 2-sided [-28.6 to 1.1]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p = 0.002, Kenward Roger; mean difference of percentage changes = -23.7, 95% CI 2-sided [-38.5 to -8.9]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p = 0.154, Kenward Roger; mean difference of percentage changes = -10.7, 95% CI 2-sided [-25.6 to 4.1]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.090, Kenward Roger; mean difference of percentage changes = -12.1, 95% CI 2-sided [-26.0 to 1.9]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p = 0.024, Kenward Roger; mean difference of percentage changes = -15.9, 95% CI 2-sided [-29.7 to -2.1]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p = 0.180, Kenward Roger; mean difference of percentage changes = -9.5, 95% CI 2-sided [-23.4 to 4.4]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.051, Kenward Roger; mean difference of percentage changes = -13.6, 95% CI 2-sided [-27.3 to 0.0]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p = 0.016, Kenward Roger; mean difference of percentage changes = -16.7, 95% CI 2-sided [-30.2 to -3.2]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p = 0.322, Kenward Roger; mean difference of percentage changes = -6.8, 95% CI 2-sided [-20.5 to 6.8]

14. Secondary Outcome: Percentage Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale (NRS) at Each Visit up to Week 24
Description: as for outcome 3
Time Frame: At baseline and Week 24
Population: ITT population: All randomized participants.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
percentage of change
  Week 1: number analyzed (Participants) | 55 | 52 | 53 | 52
  Week 1 | -9.8 (18.47) | -22.6 (21.76) | -25.5 (30.15) | -19.8 (21.16)
  Week 2: number analyzed (Participants) | 53 | 50 | 55 | 50
  Week 2 | -12.9 (23.97) | -36.9 (27.34) | -42.1 (23.91) | -37.6 (32.29)
  Week 4: number analyzed (Participants) | 52 | 50 | 51 | 49
  Week 4 | -16.3 (23.77) | -38.7 (30.25) | -51.8 (26.87) | -45.7 (32.64)
  Week 8: number analyzed (Participants) | 50 | 45 | 51 | 46
  Week 8 | -23.0 (23.88) | -48.2 (28.82) | -61.5 (24.16) | -58.0 (28.63)
  Week 12: number analyzed (Participants) | 41 | 41 | 48 | 42
  Week 12 | -28.2 (28.83) | -58.0 (28.99) | -68.7 (25.04) | -56.4 (29.81)
  Week 16: number analyzed (Participants) | 39 | 39 | 47 | 40
  Week 16 | -36.2 (30.25) | -61.4 (28.62) | -71.7 (22.53) | -63.7 (33.07)
  Week 20: number analyzed (Participants) | 34 | 37 | 41 | 36
  Week 20 | -38.0 (30.11) | -64.6 (28.62) | -69.9 (26.30) | -69.7 (28.47)
  Week 24: number analyzed (Participants) | 32 | 33 | 36 | 31
  Week 24 | -42.2 (31.66) | -65.8 (29.94) | -66.9 (38.60) | -68.2 (26.88)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 1; Test type: Superiority; p = 0.012, Kenward Roger; mean difference of percentage changes = -10.9, 95% CI 2-sided [-19.4 to -2.4]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 1; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -15.4, 95% CI 2-sided [-23.8 to -7.1]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 1; Test type: Superiority; p = 0.029, Kenward Roger; mean difference of percentage changes = -9.4, 95% CI 2-sided [-17.8 to -0.9]
Statistical Analysis 4: Comparison: Placebo vs Nemolizumab (10 mg); Week 2; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -21.8, 95% CI 2-sided [-32.0 to -11.6]
Statistical Analysis 5: Comparison: Placebo vs Nemolizumab (30 mg); Week 2; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -29.1, 95% CI 2-sided [-39.1 to -19.1]
Statistical Analysis 6: Comparison: Placebo vs Nemolizumab (90 mg); Week 2; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -23.8, 95% CI 2-sided [-34.0 to -13.6]
Statistical Analysis 7: Comparison: Placebo vs Nemolizumab (10 mg); Week 4; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -21.3, 95% CI 2-sided [-32.1 to -10.5]
Statistical Analysis 8: Comparison: Placebo vs Nemolizumab (30 mg); Week 4; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -34.8, 95% CI 2-sided [-45.5 to -24.2]
Statistical Analysis 9: Comparison: Placebo vs Nemolizumab (90 mg); Week 4; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -30.7, 95% CI 2-sided [-41.6 to -19.9]
Statistical Analysis 10: Comparison: Placebo vs Nemolizumab (10 mg); Week 8; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -22.9, 95% CI 2-sided [-33.2 to -12.6]
Statistical Analysis 11: Comparison: Placebo vs Nemolizumab (30 mg); Week 8; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -37.3, 95% CI 2-sided [-47.4 to -27.2]
Statistical Analysis 12: Comparison: Placebo vs Nemolizumab (90 mg); Week 8; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -34.1, 95% CI 2-sided [-44.4 to -23.8]
Statistical Analysis 13: Comparison: Placebo vs Nemolizumab (10 mg); Week 12; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -24.1, 95% CI 2-sided [-35.6 to -12.5]
Statistical Analysis 14: Comparison: Placebo vs Nemolizumab (30 mg); Week 12; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -38.4, 95% CI 2-sided [-49.7 to -27.2]
Statistical Analysis 15: Comparison: Placebo vs Nemolizumab (90 mg); Week 12; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -30.2, 95% CI 2-sided [-41.7 to -18.7]
Statistical Analysis 16: Comparison: Placebo vs Nemolizumab (10 mg); Week 16; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -20.9, 95% CI 2-sided [-32.8 to -8.9]
Statistical Analysis 17: Comparison: Placebo vs Nemolizumab (30 mg); Week 16; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -34.3, 95% CI 2-sided [-46.0 to -22.6]
Statistical Analysis 18: Comparison: Placebo vs Nemolizumab (90 mg); Week 16; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -28.7, 95% CI 2-sided [-40.7 to -16.8]
Statistical Analysis 19: Comparison: Placebo vs Nemolizumab (10 mg); Week 20; Test type: Superiority; p = 0.001, Kenward Roger; mean difference of percentage changes = -21.1, 95% CI 2-sided [-33.7 to -8.4]
Statistical Analysis 20: Comparison: Placebo vs Nemolizumab (30 mg); Week 20; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -29.7, 95% CI 2-sided [-42.1 to -17.3]
Statistical Analysis 21: Comparison: Placebo vs Nemolizumab (90 mg); Week 20; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -27.9, 95% CI 2-sided [-40.6 to -15.2]
Statistical Analysis 22: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p = 0.002, Kenward Roger; mean difference of percentage changes = -22.4, 95% CI 2-sided [-36.1 to -8.6]
Statistical Analysis 23: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -31.5, 95% CI 2-sided [-44.9 to -18.0]
Statistical Analysis 24: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -30.0, 95% CI 2-sided [-43.8 to -16.2]

15. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate the safety of nemolizumab in participants with moderate-to-severe AD
Time Frame: From screening to Follow-up visit (Week 32)/Early termination visit
Population: Safety population: The safety population comprised all subjects in ITT population who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 56 | 55 | 57 | 57
Participants
  Subjects with treatment-emergent SAEs | 1 | 3 | 2 | 2
  Treatment-emergent AEs (TEAE) with fatal outcome | 0 | 1 | 0 | 0
  Subjects with TEAE leading to temporary study drug | 0 | 1 | 2 | 1
  Subjects with TEAE leading to permanent study drug | 4 | 4 | 2 | 7
  Subjects with TEAE leading to study withdrawal | 0 | 3 | 2 | 3
  Subjects with at least 1 TEAE | 43 | 47 | 47 | 48
  Subjects with severe TEAEs | 6 | 3 | 5 | 2

16. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Peak Pruritus Numeric Rating Scale (NRS) at Each Visit up to Week 24
Description: Pruritus NRS is a scale to be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Time Frame: Baseline to Week 24
Population: ITT population: All randomized participants. Number of participants in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
units on a scale
  Week 1: number analyzed (Participants) | 56 | 52 | 53 | 52
  Week 1 | -0.9 (1.38) | -2.0 (1.96) | -2.3 (1.89) | -1.7 (1.66)
  Week 2: number analyzed (Participants) | 54 | 50 | 55 | 50
  Week 2 | -1.2 (1.82) | -3.1 (2.34) | -3.4 (1.96) | -3.3 (2.56)
  Week 4: number analyzed (Participants) | 55 | 50 | 53 | 50
  Week 4 | -1.4 (1.84) | -3.4 (2.62) | -4.2 (2.21) | -3.8 (2.73)
  Week 8: number analyzed (Participants) | 53 | 45 | 54 | 47
  Week 8 | -1.9 (1.94) | -4.1 (2.58) | -5.0 (2.14) | -4.7 (2.54)
  Week 12: number analyzed (Participants) | 43 | 43 | 52 | 43
  Week 12 | -2.3 (2.44) | -4.9 (2.45) | -5.6 (2.29) | -4.7 (2.66)
  Week 16: number analyzed (Participants) | 39 | 41 | 52 | 42
  Week 16 | -2.9 (2.55) | -5.2 (2.34) | -5.8 (2.25) | -5.1 (2.77)
  Week 20: number analyzed (Participants) | 36 | 40 | 47 | 38
  Week 20 | -3.1 (2.52) | -5.4 (2.61) | -5.9 (2.22) | -5.4 (2.66)
  Week 24: number analyzed (Participants) | 32 | 33 | 36 | 31
  Week 24 | -3.5 (2.65) | -5.6 (2.55) | -5.8 (2.54) | -5.5 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.0 to -1.0]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-3.8 to -1.8]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.3 to -1.3]

17. Secondary Outcome: Absolute Change From Baseline in Weekly Average of the Average Pruritus Numeric Rating Scale (NRS) at Each Visit up to Week 24
Description: Pruritus NRS is a scale to be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For average itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Time Frame: Baseline to Week 24
Population: ITT population: All randomized participants. Number of participants in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
units on a scale
  Week 1: number analyzed (Participants) | 56 | 52 | 53 | 52
  Week 1 | -0.9 (1.24) | -2.0 (1.94) | -2.3 (1.86) | -1.8 (1.64)
  Week 2: number analyzed (Participants) | 54 | 50 | 55 | 50
  Week 2 | -1.2 (1.73) | -3.1 (2.32) | -3.3 (1.89) | -3.3 (2.50)
  Week 4: number analyzed (Participants) | 55 | 50 | 53 | 50
  Week 4 | -1.5 (1.73) | -3.5 (2.47) | -4.1 (2.16) | -3.8 (2.63)
  Week 8: number analyzed (Participants) | 53 | 45 | 54 | 47
  Week 8 | -2.1 (1.95) | -4.1 (2.42) | -4.9 (2.13) | -4.7 (2.39)
  Week 12: number analyzed (Participants) | 43 | 43 | 52 | 43
  Week 12 | -2.4 (2.43) | -4.9 (2.48) | -5.5 (2.29) | -4.6 (2.50)
  Week 16: number analyzed (Participants) | 39 | 41 | 52 | 42
  Week 16 | -3.0 (2.47) | -5.3 (2.18) | -5.7 (2.19) | -5.1 (2.59)
  Week 20: number analyzed (Participants) | 36 | 40 | 47 | 38
  Week 20 | -3.3 (2.55) | -5.3 (2.47) | -5.8 (2.18) | -5.3 (2.50)
  Week 24: number analyzed (Participants) | 32 | 33 | 36 | 31
  Week 24 | -3.7 (2.59) | -5.5 (2.53) | -5.6 (2.49) | -5.2 (2.19)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.0 to -0.9]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-3.6 to -1.6]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-3.1 to -1.1]

18. Secondary Outcome: Percentage Change From Baseline in Weekly Average of the Average Pruritus Numeric Rating Scale (NRS) at Each Visit up to Week 24
Description: as for outcome 17
Time Frame: Baseline to Week 24
Population: ITT population: All randomized participants. Number of participants in this analysis
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
Number analyzed (Participants) | 57 | 55 | 57 | 57
Percentage of change
  Week 1: number analyzed (Participants) | 56 | 52 | 53 | 52
  Week 1 | -11.0 (16.33) | -24.6 (23.39) | -29.4 (28.24) | -23.2 (22.63)
  Week 2: number analyzed (Participants) | 54 | 50 | 55 | 50
  Week 2 | -14.6 (23.01) | -39.9 (29.89) | -45.2 (25.06) | -40.4 (33.77)
  Week 4: number analyzed (Participants) | 55 | 50 | 53 | 50
  Week 4 | -19.7 (22.48) | -43.5 (31.66) | -55.8 (27.60) | -48.2 (33.16)
  Week 8: number analyzed (Participants) | 53 | 45 | 54 | 47
  Week 8 | -26.9 (25.34) | -52.0 (29.50) | -65.1 (24.67) | -61.5 (28.03)
  Week 12: number analyzed (Participants) | 43 | 43 | 52 | 43
  Week 12 | -30.9 (31.63) | -61.7 (30.02) | -72.2 (25.36) | -60.1 (29.77)
  Week 16: number analyzed (Participants) | 39 | 41 | 52 | 42
  Week 16 | -40.2 (31.73) | -66.8 (27.02) | -73.9 (22.83) | -67.1 (31.64)
  Week 20: number analyzed (Participants) | 36 | 40 | 47 | 38
  Week 20 | -42.7 (32.43) | -67.5 (30.03) | -74.5 (24.85) | -70.6 (29.39)
  Week 24: number analyzed (Participants) | 32 | 33 | 36 | 31
  Week 24 | -47.7 (32.60) | -68.7 (30.60) | -69.9 (35.76) | -70.5 (26.41)
Statistical Analysis 1: Comparison: Placebo vs Nemolizumab (10 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -23.8, 95% CI 2-sided [-37.7 to -9.9]
Statistical Analysis 2: Comparison: Placebo vs Nemolizumab (30 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -31.4, 95% CI 2-sided [-45.0 to -17.7]
Statistical Analysis 3: Comparison: Placebo vs Nemolizumab (90 mg); Week 24; Test type: Superiority; p < 0.001, Kenward Roger; mean difference of percentage changes = -29.2, 95% CI 2-sided [-43.2 to -15.2]

ADVERSE EVENTS:
Time Frame: From screening to Follow-up visit (Week 32)/Early termination visit
Description: Adverse Event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product, regardless of the causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the product.
  Note: All participants in ITT population who received at least one dose of study drug were included.
Arm/Group | Placebo | Nemolizumab (10 mg) | Nemolizumab (30 mg) | Nemolizumab (90 mg)
All-Cause Mortality (participants affected / at risk) | 0/56 | 1/55 | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/55 | 2/57 | 2/57
Other Adverse Events (participants affected / at risk) | 43/56 | 47/55 | 47/57 | 47/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Nemolizumab (10 mg) (N=55) | Nemolizumab (30 mg) (N=57) | Nemolizumab (90 mg) (N=57)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Post-traumatic amnestic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | Nemolizumab (10 mg) (N=55) | Nemolizumab (30 mg) (N=57) | Nemolizumab (90 mg) (N=57)
Nasopharyngitis (Infections and infestations) | 12 | 18 | 14 | 13
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 6 | 4
Sinusitis (Infections and infestations) | 0 | 4 | 3 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 4
Oral herpes (Infections and infestations) | 1 | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 3 | 1 | 1
Rhinitis (Infections and infestations) | 3 | 0 | 3 | 1
Folliculitis (Infections and infestations) | 2 | 0 | 3 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 18 | 11 | 13 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Headache (Nervous system disorders) | 7 | 7 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information provided to the investigator and his/her staff and all data obtained through this clinical trial are confidential. The Sponsor reserves all proprietary rights. No information may be disclosed to any third party without prior written consent from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03100344/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT03100344/SAP_001.pdf